CLINICAL TRIAL: NCT04079075
Title: Multiple Interventions to Prevent Cognitive Decline
Acronym: MIND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EPIUnit_MIND_2019
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Cognitive Dysfunction; Cognition Disorders; Memory Disorders
Keywords: Correction of Hearing Impairment; Cognitive Dysfunction; Diet, Healthy; Exercise Therapy; Cognition Disorders; Neuropsychological Tests; Hearing Loss; Memory Disorders; Cognitive Remediation; Non-Randomized Controlled Trials as Topic
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders; Memory Disorders; Hearing Loss | interventions — Cognitive Training; Exercise; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-pharmacological intervention (Experimental): Non-pharmacological strategy, implemented in groups of 10 participants, over 10 consecutive months, based on five different interventions:
  cognitive training, physical activity; nutrition education; adaption to memory loss; detection and correction of hearing impairment.
  Interventions: Other: Cognitive training; Behavioral: Physical activity; Behavioral: Nutrition education; Behavioral: Adaption to memory loss; Diagnostic Test: Diagnosis of hearing impairment

INTERVENTIONS:
Other: Cognitive training — This comprises training using using the cogweb software, both in person and remotely:
  i) in person training: 30-minute sessions, supervised by a trained nurse, twice weekly .
  ii) remote training: unsupervised 30-minute sessions, to be performed at home at the participants will.
Behavioral: Physical activity — This is based on 60-minute sessions including aerobic, resistance, agility/balance and flexibility exercises, directed by a physical education teacher and supervised by a nurse, twice weekly.
Behavioral: Nutrition education — This is based on monthly 180-minute sessions, directed by a nutritionist, comprising:
  i) Presentation and discussion of healthy and easy to cook recipes by the nutritionist; ii) Preparation of healthy meals by the participants, followed by a period of social interaction between the participants while consuming the meals prepared.
Behavioral: Adaption to memory loss — This is based on monthly 30-minute sessions, directed by a psychologist or a nurse, who will provide strategies that participants may use in their daily life to cope with memory loss.
Diagnostic Test: Diagnosis of hearing impairment — Before implementing the sessions of cognitive training, physical activity, nutrition education and adaption to memory loss, an audiologist will perform an audiogram to all participants. Those with auditive performance inferior to the reference values will be referred for a medical appointment with an otolaryngologist.

SUMMARY:
The investigators aim to test the feasibility of a pragmatic non-pharmacological strategy, that may prevent cognitive decline in patients with mild cognitive impairment. This strategy is based on five different interventions: cognitive training, physical activity, nutrition education, adaption to memory loss, diagnosis and correction of hearing impairment.

A quasi-experimental study will be implemented in Porto (Portugal), including patients that fulfill all of the following criteria: a) age 18-85 years; b) Montreal Cognitive Assessment (MoCA) score greater than or equal to two standard deviations below the normative reference value for the corresponding age and education level in the Portuguese population OR diagnosis of Mild Cognitive Impairment, performed by a Neurologist, during the six previous months, considering the results of a neuropsychological battery; c) Cardiovascular Risk Factors, Aging and Dementia (CAIDE) Dementia Risk Score of at least six points. Patients who have any medical disability that contraindicates physical activity or have a lack of autonomy in daily activities will be excluded.

The program will be implemented in groups of 10 participants, over a period of 10 consecutive months.

DETAILED DESCRIPTION:
Detailed description

This is a quasi-experimental study in which the investigators aim to test the feasibility of a non-pharmacological strategy to prevent cognitive decline in patients with a diagnosis of mild cognitive impairment. This strategy is based on five different interventions:

a) Cognitive training

This comprises training using using the cogweb software, both in person and remotely:

i) in person training: 30-minute sessions, supervised by a trained nurse, twice weekly .

ii) remote training: unsupervised 30-minute sessions, to be performed at home at the participants will.

b) Physical activity This is based on 60-minute sessions including aerobic, resistance, agility/balance and flexibility exercises, directed by a physical education teacher and supervised by a nurse, twice weekly.

c) Nutrition education

This is based on monthly 180-minute sessions, directed by a nutritionist, comprising:

i) Presentation and discussion of healthy and easy to cook recipes by the nutritionist; ii) Preparation of healthy meals by the participants, followed by a period of social interaction between the participants while consuming the meals prepared.

d) Adaptation to memory loss This is based on monthly 30-minute sessions, directed by a psychologist or a nurse, who will provide strategies that participants may use in their daily life to cope with memory loss.

e) Diagnosis of hearing impairment Before implementing the sessions of cognitive training, physical activity, nutrition education and adaption to memory loss, an audiologist will perform an audiogram to all participants. Those with auditive performance inferior to the reference values will be referred for a medical appointment with an otolaryngologist.

Strategies (a),(b), (c) and (d) will be implemented over a period of 10 months, in groups of 10 participants.

ELIGIBILITY:
Inclusion criteria:

a) Age 18-85 years;

b1) Montreal Cognitive Assessment score ≥ to two standard deviations below the normative reference value for the corresponding age and education level in the Portuguese population;

OR

b2) clinical diagnosis of Mild Cognitive Impairment;

c) Cardiovascular Risk Factors, Aging and Dementia Dementia Risk Score ≥ six points.

Exclusion criteria:

1. medical disability that contraindicates physical activity;
2. lack of autonomy in daily activities.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive performance 1 | 10 months
  Variation of participant's cognitive performance assessed using the Montreal Cognitive Assessment, between the baseline assessment and the end of follow-up. This scale varies from 0 (worst cognitive performance) to 30 points (best cognitive performance).
Body mass index | 10 months
  Variation of participant's body mass index between the baseline assessment and the end of follow-up.
Adherence to the Mediterranean diet | 10 months
  Variation of participant's self-reported adherence to the Mediterranean diet, assessed using the Mediterranean food pattern (PREDIMED) scale, between the baseline assessment and the end of follow-up. This scale varies from 0 (lowest adherence to the Mediterranean diet) to 14 points (highest adherence to the Mediterranean diet). A score over 10 points indicates good adherence to the Mediterranean diet.
Number of steps | 10 months
  Variation of participant's number of steps, assessed using a portable accelerometer, between the baseline assessment and the end of follow-up.
Adherence to each intervention | 10 months
  Proportion of adherence to each intervention and component of each intervention, calculated as the number of sessions attended/total number of sessions implemented. For remote cognitive training the outcome will be the absolute number of sessions.
Dropout | 10 months
  Proportion of participants who dropped out of the study, calculated as the number of participants who dropped out after attending at least one session/total number of participants who attended at least one session.

SECONDARY OUTCOMES:
Cognitive performance 2 | 10 months
  Variation of participant's cognitive performance assessed using a neuropsychological battery, between the baseline assessment and the end of follow-up. This will be reported in the format of a Z-score, assuming positive and negative values. Higher scores indicate better cognitive performance.
Memory complaints | 10 months
  Variation of the self-reported memory complaints, assessed using the self-reported memory complaints scale, between the baseline assessment and the end of follow-up. This scale varies from 0 (best score) to 21 points (worst score). Scores over three points indicate the presence of self-reported memory complaints.
Anxiety and depression | 10 months
  Variation of the anxiety and depression scores, assessed using the Hospital Anxiety and Depression Scale (HADS), between the baseline assessment and the end of follow-up. This scale varies from 0 (best score) to 21 points (worst score).
Reported quality of life: EQ-5D scale | 10 months
  Variation of participant's quality of life, assessed using the EuroQol Group scale - 5 dimensions (EQ-5D) scale, between the baseline assessment and 10 months after the beginning of the intervention. This is assessed using two subscales: a) five multiple choice questions, with five response possibilities, which produce a score that varies from 5 (best score) to 25 points (worst score); b) visual analogic scale, that varies from 0 (worst score) to 100 (best score).
Handgrip strength | 10 months
  Variation of participant's handgrip strength, assessed using a dynamometer, between the baseline assessment and 10 months after the beginning of the intervention.
Agility 1 | 10 months
  Variation of participant's agility and balance, assessed using the Time Up and Go Test scale, between the baseline assessment and 10 months after the beginning of the intervention. This is measured in time units (seconds) and varies from 0 (best score) to infinite (worst score).
Agility 2 | 10 months
  Variation of participant's agility and balance, assessed using the One Leg Balance Test, between the baseline assessment and 10 months after the beginning of the intervention. This is measured in time units (seconds) and varies from 0 (best score) to infinite (worst score).
Time of follow-up | 10 months
  Number of days between the first and the last session attended by the participant.
Implemented sessions | 10 months
  Proportion of sessions implemented, calculated as the number of sessions that the research team was able to implement/total number of sessions planned.
Complete assessment of participants | 10 months
  For each study outcome, proportion of participants with complete information, calculated at baseline and different moments of follow-up, as the number of participants with complete information/total number of participants evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: João Firmino-Machado, MD, PhD, Principal Investigator — Instituto de Saude Publica da Universidade do Porto
Locations (1):
- Agrupamento de Centros de Saúde do Porto Ocidental, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No